CLINICAL TRIAL: NCT03777644
Title: Effect of Continuous Paravertebral Block on Postoperative Quality of Recovery After Hepatectomy
Brief Title: Continuous Paravertebral Block on Postoperative Quality of Recovery After Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: cuixulei7
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Nerve Block
MeSH Terms: interventions — Ropivacaine; Sodium Chloride; Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB + PCA (Experimental): Continuous Paravertebral block with ropivacaine and Patient-controlled analgesia with morphine
  Interventions: Procedure: Continuous Paravertebral block with ropivacaine; Drug: Patient-controlled analgesia with morphine
- placebo TPVB + PCA (Placebo Comparator): Continuous Paravertebral Block with Saline and Patient-controlled analgesia with morphine
  Interventions: Procedure: Continuous Paravertebral Block with Saline; Drug: Patient-controlled analgesia with morphine

INTERVENTIONS:
Procedure: Continuous Paravertebral block with ropivacaine — Inject local anesthetics in the T8 paravertebral space followed with catheter insertion and continuous local infusion.
  Device: Philip CX50 Ultrasound Scanner The curved (C1-5) probe of Philip CX 50 Ultrasound Scanner is used for scanning
  Device: PAJUNK Contiplex S Catheter Drug: single dose ropivacaine 0.5%ropivacaine with 1:200,000 adrenaline, 25ml in total given immediately after the correct position of the tip of the needle has been confirmed Drug: continuously infusion of ropivacaine 0.2% ropivacaine, infusion rate: 0.125ml/kg/pulse,1pulse/h given through the catheter inserted in the T8 paravertebral space following the single dose Drug: Morphine given as IPCA bolus: 2mg, lock time: 5min, 1h limitation: 8mg
  Arms: TPVB + PCA
Procedure: Continuous Paravertebral Block with Saline — Inject local anesthetics in the T8 paravertebral space followed with catheter insertion and continuous local infusion.
  Device: Philip CX50 Ultrasound Scanner The curved (C1-5) probe of Philip CX 50 Ultrasound Scanner is used for scanning
  Device: PAJUNK Contiplex S Catheter Drug: single dose saline,25ml in total given immediately after the correct position of the tip of the needle has been confirmed Drug: continuously infusion of saline 0.9% saline, infusion rate: 0.125ml/kg/pulse,1pulse/h given through the catheter inserted in the T8 paravertebral space following the single dose
  Arms: placebo TPVB + PCA
Drug: Patient-controlled analgesia with morphine — Drug: Morphine given as IPCA bolus: 2mg, lock time: 5min, 1h limitation: 8mg

SUMMARY:
Moderate to severe postoperative pain often influence patients quality of recovery after hepatectomy. Systemic opioids given with patient-controlled analgesia has been used after hepatectomy in many medical center, but the analgesic effect can be limited and undesirable side effects may bring about negative effects on patients recovery. Regional block has been proved to improve patients postoperative recovery in many kinds of surgeries.

The investigators therefore designed a prospective, randomized, subject and assessor blinded, parallel-group, placebo controlled study to test the hypothesis that continuous right thoracic paravertebral block increase patients quality of recovery score on the 7th postoperative day after hepatectomy in patients receiving i.v. patient-controlled analgesia (PCA) with morphine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo hepatectomy with J-shape subcostal incision
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
the postoperative recovery quality on postoperative day 7 | at the 7th postoperative day
  The postoperative recovery quality is evaluated with QoR-15 questionnaire. The QoR-15 is a 15-item questionnaire intended to measure QoR after anesthesia and surgery. It comprises five subscales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items) [2 Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR- 15. Anesthesiology. 2013;118(6):1332.]. Each item is scored from 0 to 10, and the possible total score ranges from 0(extremely poor quality of recovery) to 150 (excellent quality of re covery).

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 8, 24,48 hours after the surgery
  The patients evaluated their pain severity with thenumeric rating scale (NRS, 0-10),where 0 indicates no pain, and 10 indicates the most severe pain.
cumulated morphine consumption | At 8, 24,48 hours after the surgery
post operative length of stay | Up to 2 weeks
time to out-of bed activity/ambutation | Up to 2 weeks
time to resumption of bowel movement | Up to 2 weeks after surgery
the postoperative recovery quality on postoperative day 3: QoR-15 questionnaire | at the 3th postoperative day
  The postoperative recovery quality is evaluated with QoR-15 questionnaire. The QoR-15 is a 15-item questionnaire intended to measure QoR after anesthesia and surgery. It comprises five subscales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items) [2 Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR- 15. Anesthesiology. 2013;118(6):1332.]. Each item is scored from 0 to 10, and the possible total score ranges from 0(extremely poor quality of recovery) to 150 (excellent quality of re covery).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China